CLINICAL TRIAL: NCT06693440
Title: The Immune Assessment of PD-1 Antibody Therapy in Tumor - A Case-Control Study
Brief Title: The Immune Assessment of PD-1 Antibody Therapy in Tumor
Status: Recruiting | Type: Observational
Sponsor: Quanli Gao (Other Government)
Responsible Party: Sponsor-Investigator, Quanli Gao, Chief of Immunotherapy department, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Other Study IDs: HenanCH OS001
Record Dates: First submitted 2024-11-11; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Efficacy, Team; Adverse Event
Keywords: PD(L)-1 inhibitor; efficacy; adverse event
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Nivolumab; pembrolizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: PD-1 inhibitor combined therapy, 200mg, iv, q3w, 1 year for adjuvant therapy or 2 years for advanced therapy
  Interventions: Drug: PD-1 Inhibitors
- Control group: PD-1 inhibitor mono-therapy, 200mg, iv, q3w, 1 year for adjuvant therapy or 2 years for advanced therapy
  Interventions: Drug: PD-1 Inhibitors

INTERVENTIONS:
Drug: PD-1 Inhibitors — Patients received PD-1 inhibitors mono- or combined therapy in real-world clinical practice
  Other Names: Nivolumab; Pembrolizumab

SUMMARY:
This retrospective study will leverage previous immune function monitoring results in conjunction with clinical case data at this medical center.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the efficacy and safety of PD(L)-1 antibody therapy for malignant tumors in real-world settings. Treatment outcomes will be assessed according to RECIST V1.1 and iRECIST criteria, with safety graded according to CTCAE V5.0 standards. The study aims to enroll 3000 adult cancer patients treated at this center and analyze their prognosis outcomes based on previous treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Pathologically confirmed malignant tumors.
3. Complete medical records.
4. Assessable immune function test data.

Exclusion Criteria:

1. Age <18 years.
2. No confirmed tumor pathology.
3. Untraceable medical records.
4. Non-assessable immune function tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cancer
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2027-11-13 (Estimated); Study Completion 2030-11-13 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 months
  The objective response rate at 6 months
Adverse events | 1 year
  Number of participants who experienced immune-related adverse events at 1 year according to CTCAE 5.0

SECONDARY OUTCOMES:
Overall survival | 1 year
  The overall survival rate at 1 year

OTHER OUTCOMES:
Duration of response | 2 years
  The duration of response at 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Quanli Gao, Study Director — Henan Cancer Hospital
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No